CLINICAL TRIAL: NCT02006212
Title: Impact of Cerebral Monitoring on Neurologic Outcome in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Mona Momeni, MD, PhD, MD; PhD, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SARB 23th November 2013
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-01

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cadiac surgical patient; One arm (Other): All patients undergoing first or redo cardiac surgery with or without cardiopulmonary bypass necessitating general and/or local anesthesia. If they present any EEG abnormality intraoperatively an immediate cerebral CT scan will be performed and the necessary measures will be taken to reduce the neurologic damage.
  Interventions: Procedure: If any intraoperative EEG abnormality and/or asymmetry is detected a cerebral CT scan will be performed in the immediate postoperative period

INTERVENTIONS:
Procedure: If any intraoperative EEG abnormality and/or asymmetry is detected a cerebral CT scan will be performed in the immediate postoperative period

SUMMARY:
Neurologic complications after cardiac surgery range over a wide spectrum including postoperative delirium (PD), postoperative cognitive dysfunction (POCD) and cerebrovascular accidents (CVA). The incidence of these neurologic events varies depending on the type of surgery and the population studied. The incidence of PD and/or POCD is further influenced by the type of the neurologic tests used. Moreover, the timing of these tests seems to influence the results. Intraoperative cerebral monitoring is gaining importance in the anesthesia field. Recent findings have pointed out that cerebral hypoperfusion on one hand and deep levels of anesthesia on the other hand are major sources of adverse neurological outcomes, both of which can be detected with different non-invasive cerebral monitors.The present investigators are currently using the NeuroSENSE®, a processed electroencephalogram (pEEG) monitor together with cerebral near-infrared spectroscopy (NIRS) on a daily basis in every cardiac patient.

This large, prospective, observational study will investigate whether the short- and mid-term neurologic outcome of adult patients undergoing cardiac surgery are in line with observations made on the basis of the pEEG monitor NeuroSENSE® and cerebral NIRS.

DETAILED DESCRIPTION:
Whilst the incidence and the perioperative management of neurological complications after cardiac surgery may vary, they share some common risk factors for their occurrence: advanced age, cardiovascular morbidity including peripheral vascular disease, diabetes, previous stroke, preoperative cognitive impairment and dementia.As most of these factors are not modifiable at the time of surgery, conditions that can be controlled in the perioperative period should deserve more focus to prevent the occurrence of neurological problems.

Intraoperative cerebral hypoperfusion is generally accepted as a worsening factor of neurological complications.Besides hypoperfusion states, an overdose of general anesthetics is among intraoperative factors that have been evoked to influence postoperative neurological complications.

The main aim of this study is to know the incidence of POCD and PD in cardiac surgical population and to seek whether the presence and the duration of burst suppressions as detected by NeuroSENSE® on one hand and episodes of cerebral desaturation as detected by bilateral cerebral NIRS on the other hand are risk factors to develop these complications. The magnitude of burst suppression will be recorded as total Area Under the Curve (AUC) of burst suppression of each hemisphere. Cerebral desaturation is defined as AUC of 25% drop of oximetry values as compared to the preinduction values for each hemisphere. We will evaluate whether the concomitant presence of burst suppression together with cerebral oximetry desaturation can predict POCD and PD. Our study will be the first to analyze this point.

Otherwise, with this study the investigators will look for any eventual agreement between the cerebral NIRS and the NeuroSENSE® monitor in terms of detecting cerebral abnormalities. Lastly, in line with previous observations, the investigators will actively look for any intraoperative EEG abnormalities and in particular any sustained pEEG asymmetry that appears together with burst suppressions.

Although the study is observational any frontal severe EEG asymmetry together with the appearance of burst suppression will be carefully evaluated by an experienced anesthesiologist in reading and interpreting processed EEG monitor. The case will be discussed on an multidisciplinary basis and an eventual CT scan will be performed.In the absence of hemorrhage and if large cerebral vessel occlusion is identified, a catheter angiography with an eventual thrombectomy will be realized with the aim to extract the clot.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing first or redo cardiac surgery with or without cardiopulmonary bypass and with or without general anesthesia

Exclusion Criteria:

* patients sedated and/or intubated before the procedure
* patients who cannot complete the French version of Mini Mental State Examination
* patients who cannot be contacted at 6 months postoperatively

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The incidence of neurological complications is measured. Area Under the Curve (AUC) of burst suppression of each hemisphere on one hand and AUC of 25% drop of oximetry values as compared to the pre induction values on the other is measured. | Intraoperatively

SECONDARY OUTCOMES:
The concomitant existence of AUC of burst suppression with AUC of 25% drop of oximetry values are measured. | Intraoperatively
Agreement between the cerebral NIRS and the NeuroSENSE® monitor in terms of detecting BSR and Oximetry desaturation is measured. | Intraoperatively

OTHER OUTCOMES:
pEEG asymmetry together with burst suppressions are recorded. | Intraoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

REFERENCES:
- [Background] Momeni M, Baele P, Jacquet LM, Peeters A, Noirhomme P, Rubay J, Docquier MA. Detection by NeuroSENSE Cerebral Monitor of Two Major Neurologic Events During Cardiac Surgery. J Cardiothorac Vasc Anesth. 2015 Aug;29(4):1013-5. doi: 10.1053/j.jvca.2013.08.012. Epub 2013 Nov 28. No abstract available. PMID 24290745